CLINICAL TRIAL: NCT06655961
Title: The Effect of Gardening Activities on Anxiety and Psychosocial Symptoms of Hospitalized Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Elif BULUT, Research Assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOGU_HEM_EB_001
Record Dates: First submitted 2024-10-18; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Gardening; Pediatric Nursing; Activity; Psychosocial Symptoms; Anxiety; Hospital; Child; Investigation of Anxiety Levels and Psychosocial Symptoms of Children Hospitalized for Acute Diseases During Their Hospital Stay
Keywords: Hospitalized Child; Garden Activity; Pediatric Nursing; Psychosocial Symptoms; Anxiety; Mobile Garden
MeSH Terms: conditions — Motor Activity; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel group (experimental-control) randomised controlled experimental design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Children in this group will receive services within the scope of the routine treatment and nursing care protocol of the clinic during hospitalisation. No intervention will be applied to the control group of this study until the discharge process takes place. However, on the day of discharge, the children in the control group and their parents will be informed about the garden activities by the researcher. A single session gardening activity will be planned according to the request of the child and parent. During this session, children will be given the opportunity to choose a plant and a pot, and then planting, watering and creating a name card will be carried out.
  Interventions: Other: Clinical routine treatment and nursing care protocol
- Intervention Group (Experimental): Children in this group will have three sessions of gardening activities within the scope of the 'Gardening Activities Programme' during their hospitalisation. The sessions will take place only with the active participation of the child participant and the researcher (EB); there will be one child participant in each session. The duration of the sessions will be between 30-45 minutes. The sessions in the 'Garden Activities Programme' regarding the session planning of the activities to be carried out with children are as follows.
  Session 1: Pot Preparation and Plant Selection Session 2: Creating a Plant Arrangement Session 3: Care and Illustration
  Interventions: Other: Garden Activities Program

INTERVENTIONS:
Other: Garden Activities Program — When we look at the studies evaluating the effect of gardening activities on hospitalized children; it is seen that mostly children's opinions about therapeutic gardens are included and studies involving active gardening activities are limited. Shao et al. (2020) gave hospitalized children a task about garden plants and made them full this task through active participation and mobile games. However, it is seen that the gardening activity applied in this study was limited to a 5-minute task. The most important difference of our study from these studies is that a standardized gardening activity program will be applied to hospitalized children during their hospitalization and the active participation of the child will be ensured.
  Arms: Intervention Group
Other: Clinical routine treatment and nursing care protocol — Within the scope of the clinic routine treatment and nursing protocol; the decision to hospitalize the child, orientation to the clinic, execution of hospitalization paperwork, room placement, invasive intervention and treatment procedures are carried out. Treatment and care hours are revised according to individual order characteristics; 08.00-20.00, 08.00-16.00-00.00, 06.00-12.00-18.00-00.00 are planned considering the time order. 13.00-15.00 are the visiting hours. The child is not allowed to leave the clinic except for any medical purpose. No intervention will be applied to the control group of this study until the discharge process takes place.
  Arms: Control Group

SUMMARY:
The experience of hospitalization in childhood can often lead to traumatic consequences. Various practices (play, art therapy, music therapy, etc.) are used to help children cope with this process. In recent years, attention has been drawn to nature-based approaches in addition to existing practices. Within the scope of this approach, this study was planned in a parallel group (experimental-control) randomized controlled experimental design to determine the effect of garden activities on anxiety levels and psychosocial symptoms of hospitalized children aged 6-12 years. Hypotheses of the study H1: The gardening activities program applied to hospitalized children; H1a: There is an effect on children's anxiety. H1b: There is an effect on psychosocial symptoms of children. In this direction, the population of the study will consist of children between the ages of 6-12 in the children's ward of University Research and Application Hospital. The sample size determined as a result of G*power analysis was found as control (18) and intervention (18). The research will be conducted between September 2024 and June 2025. 'Child Descriptive Information Form', "Child Follow-up Form", "Child Anxiety Scale-Conditioning" and "Psychosocial Symptoms Diagnostic Scale for Hospitalized Children" will be used for data collection. The data collection process consists of three stages: pre-intervention period, intervention period and post-intervention period. Children in the intervention group will have three sessions of gardening activities within the scope of the 'Gardening Activities Program' during their hospitalization. Children in the control group will receive services within the scope of the routine treatment and nursing care protocol of the clinic during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* The age of the children is between 6-12 years old
* Hospitalization due to an acute medical diagnosis
* Hospitalization for at least 3 days
* Approval of the child's participation in the session by the responsible doctor
* The child is conscious and fully orientated
* Voluntariness of the child and parent to participate in the study

Exclusion Criteria:

* Hospitalization for more than 7 days
* No previous hospitalization experience
* High-risk drug use
* Having a chronic disease that suppresses the immune system
* Having a special condition that prevents him/her from participating in garden activities (physical, mental disability)
* Having skin conditions that prevent them from participating in garden activities
* Plant allergy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in children's anxiety as a result of the implementation of the Garden Activity Programme | Will be assessed every day from the day of admission (day 1) to the 7th day of hospitalization.
  Child Anxiety Scale-Dispositional (CAS-D): The Child Anxiety Scale-State (CAS-D) is shaped like a thermometer with a bulb at the bottom and horizontal lines with intervals going upwards. To measure the child's state anxiety, the child is asked to tick 'what he/she is feeling at the moment'. The score can range from 0-10. A high scale score indicates that the child's anxiety is increasing.
Changes in children's psychosocial symptoms as a result of the implementation of the Garden Activity Program | It will be assessed pre-intervention (1st day of hospitalization) and post-intervention (7th day of hospitalization).
  Psychosocial Symptoms Diagnostic Scale for Hospitalized Children: The scale consists of 24 items and five sub-dimensions (anxiety, hopelessness, communication difficulties, anger and aggression, regression). The scale has a 3-point likert-type scale, 'never: 0, sometimes: 1, often: 2'. The score obtained from the scale varies between 0-48. A high scale score indicates that the child hospitalized in the clinic has psychosocial problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No